CLINICAL TRIAL: NCT02730585
Title: Evaluation of the Performance of C-reactive Protein (CRP) Concentrations Variation (Delta CRP) in the Diagnosis of Acute Appendicitis in the ER
Brief Title: Diagnostic Performance of C Reactive Protein and Delta CRP in Acute Appendicitis
Acronym: dCRPappend
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: 04/2016
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Appendicitis
Keywords: C-reactive protein
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute appendicitis: all patients admitted to our hospital with a clinically suspected acute appendicitis.
  Interventions: Biological: C-reactive protein measurement

INTERVENTIONS:
Biological: C-reactive protein measurement — All patients included in this study underwent a blood sample analysis for C-reactive protein concentrations at admission and 3 hours later.

SUMMARY:
The diagnosis of acute appendicitis is difficult and despite important advances in medical sciences, detailed patient questioning and precise medical examination are the main keystones of the diagnosis of acute appendicitis and up to now, results still unsatisfactory.

DETAILED DESCRIPTION:
Acute appendicitis is the most common surgical emergency and the most common source of community-acquired intra-abdominal infections. The lack of accuracy in the diagnosis of acute appendicitis yields often to two types of outcomes: a delay in diagnosis leads to perforation and peritonitis in up to 15% of the cases and unnecessary appendectomy is associated with post-operative complications such as wound infection and adhesions. CRP is an acute phase protein that is often used by many surgeons as a diagnostic marker of acute appendicitis. During the evaluation of patients with possible appendicitis in the emergency department (ED), repeated physical examination of the abdomen may provide further information about the decision making. However, the role of repeated laboratory examinations is not proven.

The purpose of this study was to investigate whether repeated serum CRP measures could be useful to predict acute appendicitis, after 3 hours of observation, in comparison with the histopathological findings.

ELIGIBILITY:
Inclusion Criteria:

* age > 8 year old
* clinical suspicion of acute appendicitis including the presence of direct tenderness in the right lower quadrant, percussion and rebound tenderness, pyrexia, anorexia, nausea and vomiting.

Exclusion Criteria:

* patients receiving anti coagulants
* pregnant women
* patients using antibiotics during the study period.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to the Fattouma Bourguiba University hospital with an equivocal diagnosis of acute appendicitis. The clinical suspiscion of appendicitis was made based on anamnestic and physical examination findings.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Final diagnosis of acute appendicitis | 15 days from patients inclusion
  The final diagnosis of acute appendicitis was based, in operated patients, on the results of the histologic examination of the excised appendix and, in non operated patients, on the absence of acute appendicitis at the 2 weeks follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University Hospital of Monastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hallan S, Asberg A. The accuracy of C-reactive protein in diagnosing acute appendicitis--a meta-analysis. Scand J Clin Lab Invest. 1997 Aug;57(5):373-80. doi: 10.3109/00365519709084584. PMID 9279962
- [Background] Davies AH, Bernau F, Salisbury A, Souter RG. C-reactive protein in right iliac fossa pain. J R Coll Surg Edinb. 1991 Aug;36(4):242-4. PMID 1941740
- [Background] Paajanen H, Mansikka A, Laato M, Ristamaki R, Pulkki K, Kostiainen S. Novel serum inflammatory markers in acute appendicitis. Scand J Clin Lab Invest. 2002;62(8):579-84. doi: 10.1080/003655102764654312. PMID 12564616